CLINICAL TRIAL: NCT02455258
Title: Dancing for Better Aging: Evaluating the Impact of a Dance/Movement Therapy Program for Older Adults Through an Empirical Research Approach
Brief Title: Dancing for Better Aging: Evaluating the Impact of a Dance/Movement Therapy (D/MT) Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Louis Bherer, Researcher and Director of the Cognitive Health and Aging Research Lab (LESCA), Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRIUGM
Record Dates: First submitted 2015-03-31; First posted 2015-05-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Aging
Keywords: Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dance/Movement Therapy (DMT) (Experimental)
  Interventions: Other: Dance/Movement Therapy (DMT)
- Aerobics Exercise (AE) (Active Comparator)
  Interventions: Other: Aerobics Exercise (AE)
- Waiting List (No Intervention): This group is placed on a waiting list and asked to refrain from making any changes to their current lifestyle.

INTERVENTIONS:
Other: Dance/Movement Therapy (DMT) — Each DMT session follows a similar structure of Opening, Warm up, Development, Cool Down and Closure. Various themes dedicated to an aging population are addressed by the supervising dance/movement therapist through movement activities and using support material (i.e., props, music). This group is provided in a group setting of maximum 10 participants at a time and occurs 3 times per week for 1 hour each session over the course of 12 weeks.
  Arms: Dance/Movement Therapy (DMT)
Other: Aerobics Exercise (AE) — The aerobics exercise program is composed of warm up exercises followed by cardiovascular training on a recumbent bicycle. The intensity is set and progressively increased using each participants' individualized maximal aerobic power obtained in the baseline VO2 evaluation. This program respects the recommendations made by the American College of Sports Medicine and their adaptations for aging populations. Each session is supervised by a kinesiologist with 2 participants at a time. The training occurs 3 times per week for 1 hour each session over the course of 12 weeks.
  Arms: Aerobics Exercise (AE)

SUMMARY:
The aim of this study is to empirically evaluate the impact of a Dance/Movement Therapy program adapted to older adults. Participants over 60 years old are enrolled in one of three groups: Dance/Movement Therapy, Aerobic Exercise or Waiting List (control group) for 12 weeks. The training groups occur 3 times a week for 1 hour each session. Physical condition, cognitive function, general health and lifestyle, and stress hormones are assessed at baseline, after 12 weeks and after 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and older
* sedentary or moderately sedentary (less than 150 minutes of moderate to vigorous exercise per week)
* have not participated in another similar study in the last year
* have not been exposed to a dance or dance/movement therapy program in the past year
* are not in a wheelchair
* have not had surgery in the past year
* have not smoked in the past 5 years
* do not consume more than 2 glasses a day of alcohol
* are not in treatment for major depression

Exclusion Criteria:

* progressive neurological disorder
* unstable medical conditions (unstable cardio illness in the past 6 months, cardiac or thyroid troubles or pituitary gland illness)
* contraindication for moderate physical activity (major orthopaedic limitations)
* suspicion of cognitive problems (score of 24 or less on the Mini-Mental State Examination)
* large uncorrected perceptual limits
* treatment of hormone therapy
* uncontrolled hearing loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Z-score change on Cognitive Functioning | 0, 12 and 28 weeks
  Assessment of executive functions, processing speed and memory

SECONDARY OUTCOMES:
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  SF-12
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  Lubbens Social Network Scale
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  Mental Health Continuum
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  Health Promoting Lifestyle Profile
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  State-Trait Anxiety Inventory
Z-score change on Psychological Condition | 0, 12 and 28 weeks
  Depression Scale
Z-score change on Dietary Screener Questionnaire | 0,12 and 28 weeks
Z-score change on Pittsburgh Sleep Quality Index (PSQI) | 0,12 and 28 weeks
Z-score change on Brief Pain Inventory | 0, 12 and 28 weeks
Z-score change on International Consultation on Incontinence Questionnaire-Urinary Incontinence ( ICIQ-UI) | 0, 12 and 28 weeks
  Urinary Incontinence
Z-score change on Physical Functioning | 0,12 and 28 weeks
  Timed up and go
Z-score change on Physical Functioning | 0,12 and 28 weeks
  10m walk
Z-score change on Physical Functioning | 0,12 and 28 weeks
  Grip strength
Z-score change on Physical Condition | 0, 12 and 28 weeks
  VO2 peak
Z-score change on Physical Condition | 0, 12 and 28 weeks
  Bone density scanning (DEXA)
Z-score change on Physical Condition | 0, 12 and 28 weeks
  BMI
Z-score change on Physical Condition | 0, 12 and 28 weeks
  Rockport walking aerobic fitness test
Z-score change on Physical Condition | 0,12 and 28 weeks
  Anthropometric measures composite

CONTACTS AND LOCATIONS:
Locations (1):
- IUGM, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Esmail A, Vrinceanu T, Lussier M, Predovan D, Berryman N, Houle J, Karelis A, Grenier S, Minh Vu TT, Villalpando JM, Bherer L. Effects of Dance/Movement Training vs. Aerobic Exercise Training on cognition, physical fitness and quality of life in older adults: A randomized controlled trial. J Bodyw Mov Ther. 2020 Jan;24(1):212-220. doi: 10.1016/j.jbmt.2019.05.004. Epub 2019 May 7. PMID 31987547